CLINICAL TRIAL: NCT02844348
Title: Impact of Hypnosis on the Management of Chronic and Breakthrough Pain of Chronic Dialysis Patients Suffering From Arterial Disease
Brief Title: Impact of Hypnosis on Pain Management During Dialysis on Patients Suffering From Arterial Disease
Acronym: HYPNODIAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment problem
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.176; ID/RCB : 2015-A00921-48 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-05-30; First posted 2016-07-26 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Pain; Hypnosis; Chronic Dialysis; Arterial Disease
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard pain control (No Intervention): Classical pain assessment and drug treatment at each dialysis session.
- Hypnosis (Experimental): Besides the classical pain assessment and drug treatment, hypnosis sessions during 2 periods of one week of dialysis sessions.
  Interventions: Other: Hypnosis session

INTERVENTIONS:
Other: Hypnosis session
  Arms: Hypnosis

SUMMARY:
A chronic renal disease can results in the development of cardiovascular complications, including chronic arterial disease ; but a cardiovascular disease may be from a kidney malfunction that will end in end stage renal disease (ESRD). Two thirds of the chronic hemodialysis patients taken in charge in Grenoble in the last years suffered from an arterial disease at a symptomatic stage. Breakthrough pain can appear during the hemodialysis sessions. These sessions induce sudden hemodynamic changes and a peripheral vasoconstriction reaction that increases in particular all pain phenomena related to chronic low limbs ischemia. Therefore, patients have to face pain, sometimes chronic but also breakthrough pain, during the dialysis sessions, in all its dimensions.

The analgesic balance through the classical drug treatment is extremely complex, as they are both at risk of overdose and of partial effectiveness. Strict medical treatment remains unsatisfactory, as it takes into account only the expressions of symptoms during dialysis sessions, when most of the time pain is already installed and analgesic treatment is not completely effective.

The combination of classic pharmacological treatment with hypnosis, already used in other indications (chronic pain, analgesia, depression and anxiety), may mitigate the painful feeling on patients suffering from arterial disease during the dialysis sessions, with a beneficial impact on their overall quality of life. There is also evidence to suggest that hypnosis may be more effective treating neuropathic or vascular pain, those experienced by our patients, than musculoskeletal pain, like back pain.

Hypnosis is a mind-body approach focused on the subject, and not on the disease or the act of dialysis. It can be described at the same time as a modified state of consciousness and a particular intersubjective relation between a practitioner and his patient. The practice of this kind of hypnoanalgesia by the nurses is particularly relevant in hemodialysis, as the trust developed during regular chronic treatment can become an asset to shorten the induction phase and help to install this intersubjective relation.

The high incidence of this complication, the difficulties of current pain management and the impact on everyday life for the patients, justify the choice of this approach, where more further research is needed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients, requiring dialysis at least 3 times per week.
* Patients rating pain on a Visual analogue scale (VAS) > or = to 3 during hemodialysis sessions for lower limb pain related to chronic arterial disease.
* Patients affiliated to a health insurance company.
* Patients having consented to participate in the study.

Exclusion Criteria:

* Minors.
* Patients protected by law (under guardianship, deprived of liberty ...).
* Pregnant women.
* Refusal
* Patients not understanding French.
* Patients with cognitive, psychotic or behavioral disorders.
* Patients with a hearing loss limiting communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain intensity when hypnosis is applied during dialysis | up to 60 sec
  Pain is evaluate with a scale : Visual Analogue Pain Scale (VAPS) according to patients impression.

CONTACTS AND LOCATIONS:
Locations (1):
- Hemodialysis Unit University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labeeuw M, Merono Nombret A, Boyer S, Guillermin MN. Rapport du Rein Rhone Alpes Année 2012. Agence de la Biomedicine, Coordination Nationale REIN.
- [Background] Pernod G, Bosson JL, Golshayan D, Barro C, Alloatti S, Turc-Baron C, Quarello F, Jeantet A, Von Albertini B, Foret M, Lauren G, Cordonnier D, Piccoli G, Wauters JP; Diamant Alpin Collaborative Dialysis Study Group. The Diamant Alpin Dialysis cohort study: clinico-biological characteristics and cardiovascular genetic risk profile of incident patients. J Nephrol. 2004 Jan-Feb;17(1):66-75. PMID 15151261
- [Background] Rüger. Prise en charge de la douleur dans l'ischémie chronique des membres inferieurs Pain 2008 Septembre 30 139 (1) 2 : 201-208
- [Background] Santoro D, Satta E, Messina S, Costantino G, Savica V, Bellinghieri G. Pain in end-stage renal disease: a frequent and neglected clinical problem. Clin Nephrol. 2013 Jan;79 Suppl 1:S2-11. PMID 23249527
- [Background] Murtagh FE, Addington-Hall J, Higginson IJ. The prevalence of symptoms in end-stage renal disease: a systematic review. Adv Chronic Kidney Dis. 2007 Jan;14(1):82-99. doi: 10.1053/j.ackd.2006.10.001. PMID 17200048
- [Background] Bioy A. Traiter la douleur par l'hypnose. Cahier scientifique AFIDTN 2010 Dec, N°93 : 13-15.
- [Background] Le choix de l'hypnose pour soulager la douleur. Institut Upsa de la Douleur. La Douleur N°7 des recommandations à la pratique Mars 2009.
- [Background] Elkins G, Jensen MP, Patterson DR. Hypnotherapy for the management of chronic pain. Int J Clin Exp Hypn. 2007 Jul;55(3):275-87. doi: 10.1080/00207140701338621. PMID 17558718
- [Background] Dillworth T, Mendoza ME, Jensen MP. Neurophysiology of pain and hypnosis for chronic pain. Transl Behav Med. 2012 Mar;2(1):65-72. doi: 10.1007/s13142-011-0084-5. PMID 24073099
- [Background] Jensen M, Patterson DR. Hypnotic treatment of chronic pain. J Behav Med. 2006 Feb;29(1):95-124. doi: 10.1007/s10865-005-9031-6. Epub 2006 Jan 11. PMID 16404678
- [Background] Iserson KV. An hypnotic suggestion: review of hypnosis for clinical emergency care. J Emerg Med. 2014 Apr;46(4):588-96. doi: 10.1016/j.jemermed.2013.09.024. Epub 2014 Jan 25. PMID 24472351
- [Background] Kekecs Z, Varga K. Positive suggestion techniques in somatic medicine: A review of the empirical studies. Interv Med Appl Sci. 2013 Sep;5(3):101-11. doi: 10.1556/IMAS.5.2013.3.2. Epub 2013 Sep 16. PMID 24265899
- [Background] Editorial. Comfortably numb. The Association of Anaesthetists of Great Britain and Ireland 2013 ;Vol 68 : 896-898.
- [Background] Communication Journées de Néphrologie. Prouteau-Chartier M. Hypnoanalgésie en Hémodialyse chronique. Quibéron 2012
- [Background] Haute Autorite de Sante. [Management of chronic lower-limb obliterative atherosclerosis (indications for drug treatment, revascularisation and physiotherapy). Professional Guidelines Department - April 2006]. Ann Dermatol Venereol. 2007 Feb;134(2):199-206. doi: 10.1016/s0151-9638(07)91621-x. No abstract available. French. PMID 17375025
- [Background] Chauveau S. " Malades ou consommateurs ? La consommation de médicaments en France (second XXe siècle) ", Au nom du consommateur. Consommation et politique en Europe et aux Etats-Unis au XXe siècle, sous la direction de Marie Chessel, Alain Chatriot et Matthew Hilton, Paris, La Découverte, 2005, p. 182-198.
- [Background] Chan YM, Zalilah MS, Hii SZ. Determinants of compliance behaviours among patients undergoing hemodialysis in Malaysia. PLoS One. 2012;7(8):e41362. doi: 10.1371/journal.pone.0041362. Epub 2012 Aug 3. PMID 22870215
- [Background] Allen D, Wainwright M, Hutchinson T. 'Non-compliance' as illness management: Hemodialysis patients' descriptions of adversarial patient-clinician interactions. Soc Sci Med. 2011 Jul;73(1):129-34. doi: 10.1016/j.socscimed.2011.05.018. Epub 2011 May 27. PMID 21665340
- [Background] Cojan Y, Waber L, Schwartz S, Rossier L, Forster A, Vuilleumier P. The brain under self-control: modulation of inhibitory and monitoring cortical networks during hypnotic paralysis. Neuron. 2009 Jun 25;62(6):862-75. doi: 10.1016/j.neuron.2009.05.021. PMID 19555654
- [Background] Howard J. Do Bach flower remedies have a role to play in pain control? A critical analysis investigating therapeutic value beyond the placebo effect, and the potential of Bach flower remedies as a psychological method of pain relief. Complement Ther Clin Pract. 2007 Aug;13(3):174-83. doi: 10.1016/j.ctcp.2007.03.001. Epub 2007 Apr 23. PMID 17631260
- [Background] Thaler K, Kaminski A, Chapman A, Langley T, Gartlehner G. Bach Flower Remedies for psychological problems and pain: a systematic review. BMC Complement Altern Med. 2009 May 26;9:16. doi: 10.1186/1472-6882-9-16. PMID 19470153
- [Background] Rainville P. Neurophenomenologie des etats et des contenus de conscience dans l'hypnose et l'analgesie hypnotique. Théologiques, Université de Montréal, Montréal, Canada. 2004, vol. 12, no1-2, pp. 15-38.